CLINICAL TRIAL: NCT01909284
Title: Pilot Study of Efficacy and Safety of Acupuncture on Patient With Spinal Pain Due to Spondylolithesis
Brief Title: Efficacy Study of Acupuncture to Treat Spinal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Un-Suk, Noh (PhD), Department of anesthesiolgy, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIMI-13-01-20
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture & Epidural nerve block (Experimental): acupuncture plus epidural block
  Interventions: Device: Acupuncture; Procedure: Epidural nerve block
- Epidural nerve block (Active Comparator): epidural block alone
  Interventions: Procedure: Epidural nerve block

INTERVENTIONS:
Device: Acupuncture — * BL40, BL60, ST36, GB34 : bilaterally, manual acupuncture.
  * Two points on 1st bladder meridian nearest location of back pain : bilaterally, electrical acupuncture.
  Arms: Acupuncture & Epidural nerve block
Procedure: Epidural nerve block — Lumbar nerve block will be performed by using the mixture of dexamethasone (5mg) and mepivacaine (10mg).

SUMMARY:
This study is being conducted to investigate the effectiveness and safety of acupuncture for alleviating pain of spondylosis.

DETAILED DESCRIPTION:
This study is being conducted at the Daegu Catholic University Medical Center. Enrolled participants will be randomized into two groups : acupuncture treatment plus epidural block and epidural block alone.

This trial will include treatments during 3 weeks, and then follow up after 2 weeks. Participants will have acupuncture treatments of three times per week and epidural block of once per week. All examinations and treatments will be provided free of charge. Compared with epidural block group, acupuncture plus epidural block group will give more effectiveness for alleviate pain caused by lumbar spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Meyerding Grade I-II spondylolisthesis
* Low back pain of at least 1-year duration
* Follow-up possible during the clinical trial
* Written informed consent voluntarily

Exclusion Criteria:

* Cauda equina syndrome, persistently exacerbated symptoms, progressive neurologic signs (sensory or motor changes)
* Previous spine surgery
* Senile dementia, impaired cognitive function or other cerebral disease, severe psychiatric or psychological disorders
* Severe, concomitant disease (neuromuscular scoliosis, neurodegenerative disease)
* All contraindications to corticosteroid injection (e.g., insulin-dependent diabetes)
* Alcohol/drug abuse
* Significant renal or hepatic disease
* Pregnant, lactating or planning a pregnancy
* Hypersensitive reaction to acupuncture treatment
* Inability to comprehend or express oneself in the Korean language
* An individual deemed to be ineligible by a physician
* Refusal to participate in the trial or to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | Change from baseline to 5 weeks
  This outcome will measure changes in the participant's level of low back pain.

SECONDARY OUTCOMES:
Short form McGill pain questionnaire | Chagnes from baseline to 5 weeks
Oswestry Disability Index | Changes from baseline to 5 weeks
Present pain intensity(PPI) | Changes from baseline to 5 weeks
Pain vision | Chagnes from baseline to 5 weeks
  A device Pain vision Ⓡ PS-2100 calculates a "degree of pain" in cancer patients in addition to VAS

OTHER OUTCOMES:
Safety | After the initiation of acupuncture, 2 weeks, and 4 weeks
  We will confirm the safety of acupuncture by determining the red blood cell (RBC) count, hemoglobin level, platelet count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), hematocrit (Hct), total white blood cell (WBC) count, Erythrocyte Sedimentation Rate (ESR), aspartate aminotransferase (AST), alanine aminotransferase (ALT), serum urea nitrogen (BUN), creatinine level, serum sodium level, serum potassium level, and serum chloride level. All patients were evaluated 3 times, including a final follow-up visit 4 weeks after the initiation of acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-chul Seo, KMD, Ph.D., Principal Investigator — Comprehensive and Intergrative Medicine Institute; Min-Ah Gwak, KMD, Ph.D., Principal Investigator — Daegu Oriental Hospital of Daegu Haany University; Seong-Hoon Park, KMD, Principal Investigator — Comprehensive and Integrative Medicine Insitute
Locations (1):
- Daegu Catholic University Medical Center, Daegu, Kyungsangbukdo, South Korea

REFERENCES:
- [Derived] Lee HJ, Seo JC, Kwak MA, Park SH, Min BM, Cho MS, Shin I, Jung JY, Roh WS. Acupuncture for low back pain due to spondylolisthesis: study protocol for a randomized controlled pilot trial. Trials. 2014 Apr 2;15:105. doi: 10.1186/1745-6215-15-105. PMID 24693959